CLINICAL TRIAL: NCT05482048
Title: ExACT-CF: Exercise as an Airway Clearance Technique in People With Cystic Fibrosis - A Randomised Pilot Trial
Brief Title: Pilot Trial of ExACT (Exercise as Airway Clearance Therapy) for People With Cystic Fibrosis
Acronym: ExACT-CF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Royal Hospital for Children and Young People, Edinburgh (Unknown); University of Edinburgh (Other); Cystic Fibrosis Trust (Other); Department of Sport, Exercise and Rehabilitation, University of Northumbria at Newcastle (Unknown); Department of Psychology, University of Portsmouth (Unknown); Queen Elizabeth University Hospital Glasgow (Unknown); Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Zoe Saynor, Reader in Clinical Exercise Physiology, University of Portsmouth
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIHR203185
Record Dates: First submitted 2022-07-21; First posted 2022-08-01 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Two-arm randomised, pilot trial with an embedded qualitative component
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): In line with current guidelines [4], participants will continue chest physiotherapy as advised by their physiotherapist (at least one session of ACT/day) and continue to undertake exercise and physical activity at their usual levels.
- Exercise as Airway Clearance Therapy (ExACT) (Experimental): Arm-2 (ExACT): Participants will be advised to replace routine chest physiotherapy sessions with exercise combined with coughs and huffs - also referred to as forced expiratory techniques (FET) - agreed in our e-Delphi exercise REF and wider PPI discussion as possible alternatives for airway clearance. This intervention we term ExACT*.
  The undertaking of ExACT at least once per day is expected of those randomised to Arm 2.
  *Although routine chest physiotherapy is being replaced by ExACT, chest physiotherapy is permissible in the event of a chest exacerbation and a protocol deviation will be recorded.
  Interventions: Other: Exercise as Airway Clearance Therapy (ExACT)

INTERVENTIONS:
Other: Exercise as Airway Clearance Therapy (ExACT) — Arm-2 (ExACT): Participants will be advised to replace routine chest physiotherapy sessions with exercise combined with coughs and huffs - also referred to as forced expiratory techniques (FET). The undertaking of ExACT at least once per day is expected.
  Written and verbal instruction will be provided on the type, duration, frequency and intensity of exercise that is considered adequate replacement for routine chest physiotherapy. A compendium of allowable activity types, and the required times at different intensities that are considered to replace chest physiotherapy for ACT The research team will support exercise advice in line with standard care if subjects request this. The trial has no other changes to CF care. All medications, nutritional support and other treatments continue.
  Arms: Exercise as Airway Clearance Therapy (ExACT)

SUMMARY:
Cystic fibrosis (CF) is the UK s most common inherited genetic condition and affects more than 10,500 people. The disease causes problems with the movement of salt and water in the body, resulting in sticky mucus building up, mostly in the lungs and gut. Thick mucus in the airways leads to repeated infections which, over time, damage the lungs. Chest physiotherapy is prescribed to loosen and clear sticky thick mucus from the airways and so to help to reduce lung infection. Chest physiotherapy is a routine treatment to keep people with CF healthy. However, many say it is time-consuming and a burden. People with CF have asked if doing exercise could have the same effect as chest physiotherapy sessions for helping clear mucus. Exercise could be more enjoyable and less burdensome. Through a recognised priority setting partnership, the CF community recently ranked research to reduce the burden of their care and answer whether exercise can replace chest physiotherapy , as their number 1 and 7 priorities. Surveys show that many people with CF have occasionally chosen to replace chest physiotherapy with exercise for airway clearance, and we recently confirmed this through a UK-wide survey. It is not known if they would be willing to take part in research that asks some to stop chest physiotherapy and to exercise (with coughs and huffs) instead. New medicine (modulators) have recently become available for many people with CF, bringing dramatic improvements in their health. Some people who have started modulators are considering whether they can reduce or stop treatments - including chest physiotherapy. So, the effects of stopping chest physiotherapy need to be investigated and also if exercise can be used instead - this research study aims to understand this. A recent survey in people with CF, their families, physiotherapists and doctors, conducted by this research team, showed us that many consider hard exercise with coughs and huffs to be able to clear mucus from the airways. This study will recruit 50 people with CF (>12 years old) for 28-days. This study will ask half of them to continue their usual care, and half to stop chest physiotherapy and do exercise that gets them breathing deeply (with coughs and huffs) instead. This study will see if people are willing to start and continue with such a study and what they think of the study processes. It will also see how stopping chest physiotherapy and replacing it with exercise affects measurements of their lung function. The study will also involve talking with people with CF and members of their CF team to understand their experiences. This information will reveal whether a larger study can answer the question of whether certain forms of exercise can safely be used as an alternative to chest physiotherapy.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is the UK's most common inherited genetic condition and affects more than 10,500 people. People with CF have problems with the movement of salt and water in the body, which causes sticky mucus to build up, mostly in the lungs and gut. Thick mucus in the airways leads to repeated infections which may, over time, damage the lungs. All people with CF are therefore asked to use chest physiotherapy 1-2 times a day, to loosen and clear sticky thick mucus from their airways and help reduce their risk of getting a lung infection.

Chest physiotherapy is viewed as a routine treatment to keep people with CF healthy. However, many say it is time-consuming and a burden. People with CF have asked if doing exercise could have the same effect as chest physiotherapy sessions for helping clear mucus. Exercise could be more enjoyable and less burdensome and people with CF are already asked to do it regularly to stay fit and well. Surveys show that many people with CF occasionally choose to replace chest physiotherapy with exercise for airway clearance - we recently confirmed this in a UK-wide survey. It is unknown whether people with CF would be willing to take part in research that asks them to either continue with chest physiotherapy, or to stop this and do exercise (with coughs and huffs) instead.

New medicines (CFTR modulator drugs) have recently become available for many people with CF, bringing dramatic improvements in their health. Many people who have started modulators are considering whether they can reduce or stop other treatments, including chest physiotherapy. So, the effects of stopping chest physiotherapy need to be studied and research is needed to find out if exercise can be used instead - this research study aims to understand this. A recent survey in people with CF, their families, physiotherapists and doctors, undertaken by this research group, revealed that most people with CF consider exercise with coughs and huffs to be able to clear mucus from the airways in a similar manner to chest physiotherapy.

This study will recruit 50 people with CF who are older than 10 years of age for 28-days. It will randomly ask half of them to continue their usual care (chest physiotherapy), and half to stop chest physiotherapy and use exercise airway clearance therapy at least once a day instead - which will be explained to them. Briefly this will involve exercise that is ~20 minutes in duration, at a level where they must breathe deeply, used types of exercise from a list we will provide, and include assessment breaths, coughs and check huffs to help clear any sticky mucus.

This study will see if people are willing to start and continue with such a study and what they think of the study processes. It will also see how stopping chest physiotherapy and replacing it with regular exercise affects the lungs. It will also involve talking with people with CF and members of their CF team to understand their experiences of the research study. This information will reveal whether a larger study can answer the question of whether certain forms of exercise can safely be used as an alternative to chest physiotherapy and also improve what we are doing in any areas if needed.

ELIGIBILITY:
Inclusion Criteria:

* CF diagnosis based on sweat chloride >60mmol/L and CFTR genotype which includes at least one phe508del allele
* Clinically stable
* Baseline lung function (as measured by FEV1) of >40% predicted
* ≥ 10 years of age
* Established (>3 months) on Elexacaftor in combination with Tezacaftor and Ivacaftor (ETI) - Kaftrio®.
* Under the care of the paediatric centres in Southampton and Edinburgh and/or adult centres in Southampton, Edinburgh*

  *Paediatric and Adult sites in Glasgow may be utilised in event of under-recruitment to the study
* Able to cooperate with the study protocol

Exclusion Criteria:

* Considered clinically unstable by recruiting physician e.g. frequent exacerbations (>3/year in preceding 2 years), variable lung function (FEV1<40% predicted and/or excursions of >20% from baseline). Patients will not be excluded due to any pathogen as long as they are deemed clinically stable.
* Health contraindications to exercise e.g. arthritis, cardiac disease
* Not willing to give consent or to take part in the study (N.B. children will provide assent and require parent/guardian consent)
* Insufficient understanding in regard the trial - e.g. not capable of giving informed consent.
* Previously randomised into this trial
* Participation in a concurrent intervention study in the past 2 months

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants recruited into study (quantitative) | 6 months
  Number recruited and randomised 1:1 into the study

SECONDARY OUTCOMES:
Number of participants completing study (quantitative) | 28 days
  The proportion of people with CF that attend their baseline visit who also attend the Day 28 visit
Number of people completing study | 6 months
  Proportion of people with CF who complete the study and submit and necessary data
Number of people who choose intervention | 6 months
  The proportion of people with CF that would chose the intervention over usual care (chest physiotherapy) in the future
Qualitative interview data | 6 months
  Thematic analysis of semi-structured interviews of participants and healthcare professional involved with the study
Change in LCI2.5 | 28 days
  Between group differences in change in LCI2.5 from baseline to Day 28 after intervention
Change in Forced Expiratory Volume in the 1st second (FEV1) (%predicted) | 28 days
  Between group differences in change in FEV1 (%predicted) from baseline to Day 7, 14, 21 and Day 28
Change in Forced Vital Capacity (FVC) (%predicted) | 28 days
  Between group differences in change in FEV1 (%predicted) from baseline to Day 7, 14, 21 and Day 28
Rates of pulmonary exacerbations | 28 days
  Between group differences in rates of pulmonary exacerbation from baseline to Day 28
Number of adverse events | 28 days
  Between group differences in adverse events and serious adverse event rates from baseline to Day 28
Device-based physical activity (Garmin Vivosmart4 watch) | 28 days
  Between group differences in the amount/type/intensity of physical activity and exercise from baseline to Day 28
Mood | 28 days
  Between group differences in change in mood (HADS) and any change from baseline to Day 28
Quality of life (CFQ-R) | 28 days
  Between group differences in quality of life and any change from baseline to Day 28
Treatment burden | 28 days
  Between group differences in change in treatment burden (CFQ-R Treatment Burden subscale) and any change from baseline to Day 28
Habitual activity estimation scale (HAES) | 28 days
  Between group differences in change in HAES and any change from baseline to Day 28
EQ-5D-5L | 28 days
  Between group differences in change in EQ-5D-5L and any change from baseline to Day 28
Sleep | 28 days
  Between group differences in total sleep time and any change from baseline to Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Zoe Saynor, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Urquhart DS, Taylor E, Cunningham S, Lewis S, Neilson AR, Soilemezi D, Ensor H, Vogiatzis I, Allen LJ, Saynor ZL; ExACT-CF Study Group. Safety, feasibility and efficacy of exercise as an airway clearance technique in cystic fibrosis: a randomised pilot feasibility trial. Thorax. 2025 Oct 1:thorax-2025-223080. doi: 10.1136/thorax-2025-223080. Online ahead of print. PMID 41033804
- [Derived] Urquhart DS, Cunningham S, Taylor E, Vogiatzis I, Allen L, Lewis S, Neilson AR, Soilemezi D, Akooji N, Saynor ZL. Exercise as an Airway Clearance Technique in people with Cystic Fibrosis (ExACT-CF): rationale and study protocol for a randomised pilot trial. NIHR Open Res. 2022 Dec 19;2:64. doi: 10.3310/nihropenres.13347.1. eCollection 2022. PMID 37881306